CLINICAL TRIAL: NCT06401629
Title: The UPDATE-GDM Study: OUtcomes After NPRP anD ConventionAl CriTEria for GDM Diagnosis: A Pragmatic Randomised Trial
Brief Title: Outcomes After Unified Versus Standard GDM Diagnosis
Acronym: UPDATE-GDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Suhail A. Doi, Principal Investigator, Qatar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ARG02-0403-240134
Record Dates: First submitted 2024-05-01; First posted 2024-05-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gestational Diabetes; Diagnosis; Pregnancy
Keywords: Gestational Diabetes Mellitus; IADPSG; NPRP; Obesity; Dysglycemia; High-risk Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Disease; Obesity

STUDY DESIGN:
Intervention Model Description: This study will be designed as a multicentre, two-arm, parallel, pragmatic, randomized controlled trial conducted at two participating hospitals in Qatar. This design allows for an assessment of interventions in real-world settings and offers practical insights into the clinical utility of different diagnostic criteria. All pregnancies will be randomly assigned to the NPRP or IADPSG approach (1:1 ratio) at their first prenatal visit using an electronically generated random assignment procedure; this assignment will be provided to the lab within CERNER at the time of reporting GDM screening results (typically done at 24-28 weeks' gestation). If screening was ordered more than once, the same assigned result type will be presented to providers each time.
Who Masked: Participant, Outcomes Assessor
Masking Description: Owing to the pragmatic trial design, providers will not be blinded to randomization. All outcome assessors will be blinded until randomization is completed for all patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- National Priorities Research Program (NPRP) diagnostic criterion (Experimental): Interventional diagnostic strategy
  Interventions: Diagnostic Test: NPRP criteria
- International Association of Diabetes and Pregnancy Study Groups (IADPSG) diagnostic criterion (Active Comparator): Control diagnostic strategy
  Interventions: Diagnostic Test: IADPSG criteria

INTERVENTIONS:
Diagnostic Test: NPRP criteria — Under the NPRP criterion, the plasma glucose level at each time point (TP1, TP2, and TP3) is multiplied by its weight (Doi et al. 2022), and the sum of these products yields the unified Doi's Weighted Average Glucose (dwAG) value for each woman. The dwAG is then categorized into four groups: a dwAG of 6.8 or lower, >6.8 to ≤7.5, >7.5 to ≤8.6, and above 8.6 mmol/L, indicating normal gestational glycemia (NGG), impaired gestational glycemia (IGG), gestational diabetes mellitus (GDM), and high-risk gestational diabetes mellitus (hGDM), respectively (Doi et al. 2022).
  Arms: National Priorities Research Program (NPRP) diagnostic criterion
Diagnostic Test: IADPSG criteria — The IADPSG criteria define GDM as any one of the three-time points above specific thresholds: the time point prior to glucose ingestion (TP1) is considered abnormal when the fasting plasma glucose (FPG) value is ≥ 5.1 mmol/L, the 1-hour time-point after glucose ingestion (TP2) is considered abnormal when the value is ≥ 10 mmol/L, and the 2-hour time-point after glucose ingestion (TP3) is considered abnormal when the Post-Load Plasma Glucose levels are ≥ 8.5 mmol/L (Metzger et al. 2010). Put simply, meeting any one of these cut-offs results in a GDM diagnosis, regardless of whether the other time points show normal values or not (Metzger et al. 2010).
  Arms: International Association of Diabetes and Pregnancy Study Groups (IADPSG) diagnostic criterion

SUMMARY:
Gestational diabetes mellitus (GDM) is a condition that can affect pregnant women during pregnancy and may cause complications for the mother and the baby. Therefore, early and accurate detection is necessary to provide the woman and the baby with better health outcomes. Currently, the most commonly used criteria to detect GDM is the International Association of Diabetes and Pregnancy Study Groups (IADPSG) criterion. However, there is a suggestion that it results in over-diagnosis of GDM, and newer methods of diagnosis have been proposed. One such proposal is to have more than a binary outcome of assessment of dysglycemia in pregnancy. The investigator group created this criterion known as the National Priorities Research Program (NPRP) criterion. This clinical trial compares the IADPSG to the NPRP criteria in pregnant women in Qatar to determine if this newer method mitigates overdiagnosis and more accurately identifies women at risk of complications.

DETAILED DESCRIPTION:
This research project explores a crucial aspect of maternal and fetal health: the diagnosis of gestational diabetes mellitus (GDM), a condition that poses risks to both pregnant women and the babies. Gestational diabetes is a condition that can develop during pregnancy, characterized by dysglycemia and associated risks of complications such as pre-eclampsia, cesarean delivery, and macrosomia. For the baby, it raises the risk of developing obesity, type 2 diabetes later in life, and metabolic syndrome. Therefore, early and accurate diagnosis is paramount to manage and mitigate these risks. The IADPSG (International Association of Diabetes and Pregnancy Study Groups) criteria, the current standard for GDM diagnosis, has been widely adopted due to its putative sensitivity in detecting GDM and potential for reducing GDM-related complications. However, this method is not without its limitations, including the risk of over- or under-diagnosis of GDM. This project will investigate the efficacy of an alternative diagnostic method, the National Priorities Research Program (NPRP) criteria, against the conventional IADPSG criteria, diagnosis usually being undertaken between the 24th and 28th weeks of pregnancy. The NPRP criteria are based on a unified assessment of the oral glucose tolerance test (GTT), which could offer a four-level classification of dysglycemia in pregnancy as opposed to the binary diagnosis by the IADPSG criteria, thus having the added benefit of glycemic risk stratification during pregnancy. By comparing the outcomes of pregnancies diagnosed using the NPRP criteria against those diagnosed using the IADPSG criteria, the investigators aim to assess whether the NPRP criteria can provide improved outcomes (Bashir et al. 2021) in terms of maternal and fetal health through better informed GDM-related decision-making. In addition, this study proposes the NPRP criteria as potentially able to mitigate over- and under-diagnosis of GDM. This study will employ a parallel-group, prospective, randomized, pragmatic, controlled trial design and the study investigators will work closely with a cohort of pregnant women throughout pregnancy, employing both diagnostic methods to evaluate their impact on the health of the mother and the baby. The evaluation will not only focus on the immediate outcomes during pregnancy but will also aim to follow up on longer-term metabolic health implications for both mother and child post-delivery after the trial is completed and if the participant consents to such additional follow-up. The significance of this research lies in its potential to transform the current practices in GDM diagnosis, by offering evidence on the effectiveness and benefits of the NPRP criteria, thus paving the way for a shift towards a more patient-centered approach to the diagnosis of gestational diabetes. Determining if the NPRP criteria can lead to better health outcomes for mothers and babies can have profound implications for maternal and child health. Improved diagnostic methods could lead to more timely interventions, reducing the prevalence of complications associated with gestational diabetes and improving the quality of life for countless families. Through this study, the investigators hope to make a significant contribution to the well-being of pregnant women and babies, ensuring a healthier start for the next generation.

ELIGIBILITY:
Inclusion Criteria:

* This will include broad eligibility criteria of age 18-45 years with or without risk factors at first antenatal care (ANC) visit who are willing to undergo testing at 24-28 weeks and able to provide informed consent.

Exclusion Criteria:

* a multiple pregnancy at the time of screening, pre-existing diabetes (T1DM, T2DM)
* any medical condition affecting glucose metabolism or the results of the GTT (e.g., Cushing's syndrome, bariatric surgery history)
* known history of major conditions that could interfere with the study or pregnancy outcomes (e.g., severe liver, renal or cardiovascular disorders, chronic infections).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2650 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
large for gestational age (LGA) | Through pregnancy completion, an average of 9 months
  infants who weigh > 90th percentile for gestational age

SECONDARY OUTCOMES:
Average plasma glucose | Through pregnancy completion, an average of 9 months
  Report: Group mean and standard deviation (SD); for both pre-prandial and 2 hour postprandial glucose
Glycemic targets unmet | Through pregnancy completion, an average of 9 months
  Reports: Number with any of the following: Need to move to insulin; readmission for poor glycemic control; intervention targets unmet
Adverse events related to treatment | Through pregnancy completion, an average of 9 months
  Report: Number (by group) reporting any GI or systemic adverse effects and split by:
  1. Maternal hypoglycemia (glucose < 4 mmol/L or who received inter-venous glucose rescue)
  2. Others (excluding hypoglycemia)
Total weight gain in pregnancy (kg) | Through pregnancy completion, an average of 9 months
  Report: Group means and SD of total weight gained during pregnancy
Birth weight (newborn's weight at birth) | Through pregnancy completion, an average of 9 months
  Report: Numbers (by group) with LGA as well as group means and SD of continuous birth weight
Hypoglycemia within 1 hour of birth | Through pregnancy completion, an average of 9 months
  Report: Number (by group) with hypoglycemia (<=1.65 mmol/L)
Neonatal composite morbidity and mortality outcome | Through pregnancy completion, an average of 9 months
  Report: number (by group) of any neonatal death, stillbirth, or neonatal intensive care unit (NICU) admission and also split by:
  1. NICU admission > 24 hours
  2. Neonatal death (within 28 days of birth)
  3. Stillbirth
Assisted labor/delivery (including cesarean) | Through pregnancy completion, an average of 9 months
  Report: Number (by group) of all assisted deliveries as well as split by:
  1. Non-cesarean: any of induction/augmentation/vacuum extraction/operative vaginal delivery etc.
  2. Elective/Emergency Cesarean Section
  3. Primary/repeated Cesarean Section
Preterm delivery | Through pregnancy completion, an average of 9 months
  Report: Number (by group) with delivery at <37 weeks of gestation
Peripartum infection | Through pregnancy completion, an average of 9 months
  Report: Number (by group) of any of chorioamnionitis, urinary tract infections (UTI) or any other maternal infections
Pregnancy induced hypertension (PIH) or pre-eclampsia/ eclampsia | Through pregnancy completion, an average of 9 months
  Report: Number (by group) of all PIH as well as split by
  1. Eclampsia/pre-eclampsia
  2. Other PIH

OTHER OUTCOMES:
Additional composite outcome | Through pregnancy completion, an average of 9 months
  A composite of PIH, preterm delivery, LGA, NICU admission for >24h, and stillbirth after 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Suhail A. Doi, MBBS, PhD, Principal Investigator — Qatar University

IPD SHARING:
Plan to Share IPD: No
No plans at this point.

REFERENCES:
- [Background] Doi SAR, Bashir M, Sheehan MT, Onitilo AA, Chivese T, Ibrahim IM, Beer SF, Furuya-Kanamori L, Abou-Samra AB, McIntyre HD. Unifying the diagnosis of gestational diabetes mellitus: Introducing the NPRP criteria. Prim Care Diabetes. 2022 Feb;16(1):96-101. doi: 10.1016/j.pcd.2021.08.006. Epub 2021 Aug 19. PMID 34419366
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Bashir M, Syed A, Furuya-Kanamori L, Musa OAH, Mohamed AM, Skarulis M, Thalib L, Konje JC, Abou-Samra AB, Doi SAR. Core outcomes in gestational diabetes for treatment trials: The Gestational Metabolic Group treatment set. Obes Sci Pract. 2021 Feb 3;7(3):251-259. doi: 10.1002/osp4.480. eCollection 2021 Jun. PMID 34123392